CLINICAL TRIAL: NCT03038412
Title: Clinical Detection and Quantification of Caries and Dental Plaque Based on Auto-fluorescence Imaging System: An Observational Study
Brief Title: Clinical Assessment of Caries and Dental Plaque Based on Auto-fluorescence Imaging System
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Hui Chen (Other)
Responsible Party: Sponsor-Investigator, Hui Chen, Professor, The Dental Hospital of Zhejiang University School of Medicine
Organization: The Dental Hospital of Zhejiang University School of Medicine (Other)
Other Study IDs: DHZhejiangU1
Record Dates: First submitted 2017-01-30; First posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2017-01

CONDITIONS: Dental Caries (Diagnosis); Dental Plaque; Optical Imaging
MeSH Terms: conditions — Dental Caries; Disease; Dental Plaque

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional

SUMMARY:
The purpose of this study was to evaluate the applicability of auto-fluorescence imaging system to detect and quantify caries and dental plaque. Participants were advised to rinse their mouth with distilled water to exclude any chance of fluorescence from food debris. A well trained physicist majored in optical spectroscopy captured auto-fluorescence images of buccal aspects of two maxillary central incisors and occlusal aspects of four first molars from each patient in a dark room. Then they chewed a disclosing agent to assess the Quigley Hein plaque index modified by Turesky of each tooth. Furthermore, participants were also required to brush their teeth for 3min, then International Caries Detection and Assessment System（ICDAS）codes of relevant teeth to evaluate degrees of caries were recorded by an experienced dentist using a mouth mirror and explorer. The Spearman rank correlation coefficient between colorimetric parameters of fluorescence image and the plaque index and ICDAS code were calculated to evaluate the sensitivity and specificity of auto-fluorescence imaging system.

ELIGIBILITY:
Inclusion Criteria:

Subjects were required to:

* 1. have two maxillary central incisors and four first molars in mouth;
* 2. have caries in their mouth or have a high risk to get caries and need to be treated by dentists ;
* 3. sign informed consent form.

Exclusion Criteria:

* 1.two incisors and four first molars of participants ever received endodontics treatment;
* 2. history of antibiotics, mouthwashes, or any periodontal treatment during the last 3 months;
* 3.with calculus and cementum exposed in tooth cervical;
* 4. active systemic disease;
* 5. physical or mental disability;
* 6. pregnant or lactating.

Ages: 18 Years to 54 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consisted of 60 patients are from the Affiliated Stomatology Hospital of Medical College, Zhejiang University. They have caries in their mouth and need to be treated by dentists with filling cavity. Two maxillary central incisors and four first molars exist in each patient.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-05 (Actual); Primary Completion 2017-05 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Auto-fluorescence image assessment | 1 week after image collection
  Colorimetric parameters of auto-fluorescence images of buccal aspects of two maxillary central incisors and occlusal aspects of four first molars from each patient were calculated to get the Percentage Plaque Index (PPI). PPI is defined as the ratio between area of dental plaque on teeth and the whole teeth area.
The Quigley Hein plaque index modified by Turesky | right after disclosing
  After disclosing dental plaque, plaque index was evaluated as following scoring system:0 no plaque;
  1. separate flecks of plaque at the cervical margin of the margin of the tooth;
  2. a thin continuous band of plaque (up to 1 mm) at the cervical margin;
  3. a band of plaque wider than 1 mm but covering less than (1/3)rd of crown;
  4. plaque covering at least (1/3)rd but less than (2/3)rd of the crown;
  5. plaque covering (2/3)rd or more of the crown
ICDAS scoring results | right after oral detection
  After brushing teeth, ICDAS codes were recorded by an experienced dentist using a mouth mirror and explorer:0 sound；
  1. first visual change in enamel;
  2. distinct visual change in enamel;
  3. localized enamel breakdown;
  4. underlying dentine shadow;
  5. distinct cavity with visible dentine;
  6. extensive cavity within visible dentine.

CONTACTS AND LOCATIONS:
Overall Officials: Hui Chen, Study Chair — Affiliated Hospital of Stomatology, College of Medicine, Zhejiang University

IPD SHARING:
Plan to Share IPD: Undecided